CLINICAL TRIAL: NCT01852370
Title: Bilateral Orthotopic Lung Transplant in Tandem With CD3+ and CD19+ Cell Depleted Bone Marrow Transplant From Partially HLA-Matched Cadaveric Donors
Brief Title: Sequential Cadaveric Lung and Bone Marrow Transplant for Immune Deficiency Diseases
Acronym: BOLT+BMT
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Paul Szabolcs (Other)
Responsible Party: Sponsor-Investigator, Paul Szabolcs, Chief, Division of Blood and Marrow Transplant, Children's Hospital of Pittsburgh of UPMC, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19090108
Record Dates: First submitted 2013-04-26; First posted 2013-05-13 (Estimated); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Severe Combined Immunodeficiency (SCID); Immunodeficiency With Predominant T-cell Defect, Unspecified; Severe Chronic Neutropenia; Chronic Granulomatous Disease (CGD); Hyper IgE Syndromes; Hyper IgM Deficiencies; Wiskott-Aldrich Syndrome; Mendelian Susceptibility to Mycobacterial Disease; Common Variable Immune Deficiency (CVID)
Keywords: Lung transplantation; Bone Marrow Transplantation; Unrelated Donor; Cadaveric Donor; Deceased Donor; HLA-mismatch; BOLT; BMT; HSCT
MeSH Terms: conditions — Severe Combined Immunodeficiency; Neutropenia, severe chronic; Granulomatous Disease, Chronic; Job Syndrome; Wiskott-Aldrich Syndrome; Common Variable Immunodeficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BOLT+BMT (Experimental): All patients will receive a double lung transplant followed by a hematopoietic stem cell transplant. The lungs and stem cells are from the same partially HLA-matched cadaveric donor. Prior to transplantation, the marrow will be negatively selected for CD3/CD19 using a CliniMACS® depletion device.
  Interventions: Biological: CD3/CD19 negative allogeneic hematopoietic stem cells

INTERVENTIONS:
Biological: CD3/CD19 negative allogeneic hematopoietic stem cells — Negative selection for CD3/CD19 will be performed on a CliniMACS® depletion device within 36 hours of collection and given at time no less than 8 weeks post lung transplant.

SUMMARY:
The purpose of this study is to determine whether bilateral orthotopic lung transplantation (BOLT) followed by cadaveric partially-matched hematopoietic stem cell transplantation (HSCT) is safe and effective for patients aged 5-45 years with primary immunodeficiency (PID) and end-stage lung disease.

DETAILED DESCRIPTION:
This is an original IND for an investigator initiated phase I/II study. The primary purpose of the study is to evaluate the safety and efficacy of performing bilateral orthotopic lung transplantation (BOLT) followed by cadaveric, partially HLA-matched CD3+/CD19+-depleted hematopoietic stem cell transplantation (HSCT) from the same donor for patients with primary immunodeficiency diseases (PID) and end-stage lung disease. For many patients with primary immunodeficiencies, HSCT is a curative, life-saving therapy, resulting in restoration of function in the immune system. Patients with primary immunodeficiencies often develop pulmonary complications as a result of chronic or recurrent infections, making them ineligible for HSCT due to the high risk of mortality and pulmonary complications. Lung transplant prior to HSCT would allow for restoration of pulmonary function prior to HSCT, allowing PID patients to proceed to HSCT, which would be curative for the patient's underlying immunodeficiency. As a secondary aim after successful engraftment with donor bone marrow, there is realistic hope for tolerating planned withdrawal of immunosuppression achieving eventual freedom from all immunosuppressive drugs and attaining a tolerant state.

ELIGIBILITY:
Inclusion Criteria

1. Subject and/or parent guardian must be able to understand and provide informed consent.
2. Male or female, 5 through 45 years old, inclusive, at the time of informed consent.
3. Patients must have evidence of an underlying primary immunodeficiency for which BMT is clinically indicated.

   Examples of such diseases include, but are not limited to:
   * Severe Combined Immunodeficiency
   * Combined immunodeficiency with defects in T-cell-mediated immunity, including Omenn syndrome and DiGeorge Syndrome
   * Severe Chronic Neutropenia
   * Chronic Granulomatous Disease
   * Hyper IgE Syndrome or Job Syndrome
   * CD40 or CD40L deficiency
   * Wiskott-Aldrich Syndrome
   * Mendelian Susceptibility to Mycobacterial Disease [6]
   * GATA2 Associated Immunodeficiency NOTE: A genetic diagnosis is recommended, but not required.
4. Patients must have evidence of end-stage lung disease and be candidates for bilateral orthotopic lung transplant as determined by the lung transplant team.
5. GFR ≥ 50 mL/min/1.73 m2.
6. AST, ALT ≤ 4x upper limit of normal, total bilirubin ≤ 2.5 mg/dL, normal INR.
7. Cardiac ejection fraction ≥ 40% or shortening fraction ≥26%.
8. Negative pregnancy test for females >10 years old or who have reached menarche, unless surgically sterilized.
9. All females of childbearing potential and sexually active males must agree to use a FDA approved method of birth control for up to 24 months after BMT or for as long as they are taking any medication that may harm a pregnancy, an unborn child or may cause birth defect.
10. Subject and/or parent guardian will also be counseled regarding the potential risks of infertility following BMT and advised to discuss sperm banking or oocyte harvesting.

Exclusion Criteria

Individuals who meet any of these criteria are not eligible for this study:

1. Inability or unwillingness of a participant to give written informed consent or comply with study protocol.
2. Patients who have underlying malignant conditions.
3. Patients who have non-malignant conditions not requiring hematopoietic stem cell transplantation.
4. HIV positive by serology or PCR, HTLV positive by serology.
5. Females who are pregnant or who are lactating.
6. Allergy to DMSO or any other ingredient used in the manufacturing of the stem cell product.
7. Uncontrolled pulmonary infection, as determined by radiographic findings and/or significant clinical deterioration. NOTE: Pulmonary colonization with multiple organisms is common, and will not be considered an exclusion criterion.
8. Uncontrolled systemic infection, as determined by the appropriate confirmatory testing e.g. blood cultures, PCR testing, etc.
9. Recent recipient of any licensed or investigational live attenuated vaccine(s) within 4 weeks of transplant.
10. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

Eligibility Criteria to proceed to Bone Marrow Transplant

1. GFR ≥ 50 mL/min/1.73 m2.
2. AST, ALT ≤ 4x upper limit of normal, total bilirubin ≤ 2.5 mg/dL.
3. Cardiac ejection fraction ≥ 40% or shortening fraction of at least 26%.
4. HIV negative by serology and PCR.
5. HTLV serology negative.
6. FVC and FEV1 ≥40% predicted for age and SpO2 of >90% at rest on room air AND with clearance by the lung transplant team.
7. Absence of uncontrolled infection as determined by positive blood cultures and radiographic progression of previous sites in particular pulmonary densities during the past 2 weeks prior to chemotherapy.
8. Absence of clinically significant Acute Cellular Rejection (A2-A4 and/or B2R rejection).

Ages: 5 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Estimated)
Dates: Start 2013-06-20 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Safety: Death | Up to 2 years post stem cell transplant
  How many, if any, patients die.
Safety: Engraftment syndrome | Up to 2 years post stem cell transplant
  How many, if any, patients develop engraftment syndrome.
Safety: Engraftment failure | Up to 2 years post stem cell transplant
  How many patients, if any, develop engraftment failure.
Safety: Rituximab | Up to 2 years post stem cell transplant
  The number of grade 4 and 5 events potentially related to rituximab.
Efficacy: BOS score | 1 year post stem cell transplant
  Bronchiolitis Obliterans Syndrome (BOS) score for all patients who receive both lungs and stem cell transplants.
Efficacy: T-cell chimerism | 1 year post stem cell transplant
  The number of patients who have ≥ 25% donor T-cell chimerism.
Efficacy: Myeloid chimerism | 1 year post stem cell transplant
  The number of patients with myeloid disorders (e.g. CGD) who attain ≥ 10% myeloid chimerism.
Efficacy: B-cell chimerism | 1 year post stem cell transplant
  The number of patients with B-cell disorders who attain ≥ 10% B-cell chimerism.

SECONDARY OUTCOMES:
Feasibility of meeting BMT eligibility critieria | Up to 2 years post stem cell transplant
  The number of patients who are able to proceed to BMT within 6 months following lung transplant.
Tolerance | Up to 2 years post stem cell transplant
  Development of tolerance to both the host and pulmonary graft.
Long-term complications | Up to 2 years post stem cell transplant
  Long-term complications of combined solid organ and BMT.
Graft failure | Up to 2 years post stem cell transplant
  The number of patients who develop graft failure.
Acute cellular rejection | Up to 2 years post stem cell transplant
  The number of patients who develop acute cellular rejection.
Acute graft-versus-host disease (GVHD) | Up to 2 years post stem cell transplant
  The number of patient who develop acute graft-versus-host disease (GVHD).
Chronic graft-versus-host disease (GVHD) | Up to 2 years post stem cell transplant
  The number of patient who develop chronic graft-versus-host disease (GVHD).
Ability to withdraw immunosuppression | 1 year post stem cell transplant
  The number of patients who are able to start immunosuppression withdrawal.
Time to withdraw immunosuppression | Up to 2 years post stem cell transplant
  Time from BMT to withdrawal of immunosuppression.
Pathogen-specific immunity | Up to 2 years post stem cell transplant
  Time from BMT to independence from treatment dose antimicrobial drugs.
Lymphocyte count - for T-cell lymphopenias | 1 year post stem cell transplant
  The number of patients who are able to achieve an age adjusted, low limit normal range lymphocyte count.
Chronic lung allograft dysfunction | 1 year post lung transplant
  The number of patients who develop chronic lung allograft dysfunction post-lung transplant for all subjects, lung only and lung+stem cell transplant.
Allograft failure | 1 year post lung transplant
  The number of patients who develop allograft failure post-lung transplant for all subjects, lung only and lung+stem cell transplant.
Rituximab related adverse events | From the time of the first dose of rituximab up to the start of BMT conditioning.
  The number of grade 4 or 5 adverse events possibly related to the use of rituximab.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Szabolcs, MD, Principal Investigator — Division of BMT and Cellular Therapy, Children's Hospital of Pittsburgh of UPMC
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No